CLINICAL TRIAL: NCT01062763
Title: South Danish Hypertension and Diabetes Study
Brief Title: The Effect of Spironolactone on Blood Pressure in Type-2 Diabetics With Resistant Hypertension
Acronym: SDHDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ib Abildgaard Jacobsen (Other)
Responsible Party: Sponsor-Investigator, Ib Abildgaard Jacobsen, Consultant physician, associate professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT 2009-017033-22; 2009-017033-22 (EudraCT Number)
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Arterial Hypertension; Hypertension, Resistant to Conventional Therapy; Diabetes Mellitus
Keywords: hypertension; spironolactone; antihypertensive treatment; Type-2 diabetes
MeSH Terms: conditions — Hypertension; Hypertension Resistant to Conventional Therapy; Diabetes Mellitus | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- addition of spironolactone (Experimental): spironolactone is added to previous antihypertensive treatment
  Interventions: Drug: spironolactone
- Placebo (Placebo Comparator): Addition of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: spironolactone — 25 to 50 mg once daily
  Arms: addition of spironolactone
Drug: placebo — addition of placebo 1 to 2 tablets daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to estimate the effect of spironolactone on blood pressure resistant to therapy in type-2 diabetics.

DETAILED DESCRIPTION:
The primary object of the study is to estimate the effect of addition of low dose spironolactone to antihypertensive treatment with at least three antihypertensive drugs in patients with type-2 diabetes and blood pressure over 130/80 mmHg.

Secondary aims are to estimate how many of these patients have their blood pressure controlled by the addition of spironolactone, to investigate whether the addition of spironolactone affects insulin sensitivity and urinary protein secretion and to estimate the incidence of adverse effects of the aldosterone antagonist.

ELIGIBILITY:
Inclusion Criteria:

* Age < 75 years
* Type-2 diabetes
* Therapy resistant hypertension (by ABPM)
* Treatment with at least 3 antihypertensives

Exclusion Criteria:

* HbA1c > 10.0
* BP > 180/110 mmHg
* Secondary hypertension
* Intolerance to spironolactone
* Permanent treatment with nonsteroidal antiinflammatory drugs or systemic glucocorticoids
* Total cholesterol 10 mmol/l
* New York Heart Association class III and IV
* Pregnancy or planned pregnancy
* Psychiatric disease
* Malignant disease
* Insufficient adherence

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ib A Jacobsen, DMSc, Principal Investigator — Odense University Hospital

REFERENCES:
- [Background] Elliott HL, Elawad M, Wilkinson R, Singh SP. Persistence of antihypertensive efficacy after missed doses: comparison of amlodipine and nifedipine gastrointestinal therapeutic system. J Hypertens. 2002 Feb;20(2):333-8. doi: 10.1097/00004872-200202000-00025. PMID 11821720
- [Background] Nishizaka MK, Zaman MA, Calhoun DA. Efficacy of low-dose spironolactone in subjects with resistant hypertension. Am J Hypertens. 2003 Nov;16(11 Pt 1):925-30. doi: 10.1016/s0895-7061(03)01032-x. PMID 14573330
- [Background] Sharabi Y, Adler E, Shamis A, Nussinovitch N, Markovitz A, Grossman E. Efficacy of add-on aldosterone receptor blocker in uncontrolled hypertension. Am J Hypertens. 2006 Jul;19(7):750-5. doi: 10.1016/j.amjhyper.2005.11.016. PMID 16814132
- [Background] Chapman N, Dobson J, Wilson S, Dahlof B, Sever PS, Wedel H, Poulter NR; Anglo-Scandinavian Cardiac Outcomes Trial Investigators. Effect of spironolactone on blood pressure in subjects with resistant hypertension. Hypertension. 2007 Apr;49(4):839-45. doi: 10.1161/01.HYP.0000259805.18468.8c. Epub 2007 Feb 19. PMID 17309946
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- [Derived] Oxlund CS, Cangemi C, Henriksen JE, Jacobsen IA, Gram J, Schousboe K, Tarnow L, Argraves WS, Rasmussen LM. Low-dose spironolactone reduces plasma fibulin-1 levels in patients with type 2 diabetes and resistant hypertension. J Hum Hypertens. 2015 Jan;29(1):28-32. doi: 10.1038/jhh.2014.27. Epub 2014 Apr 17. PMID 24739800

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from outpatient clinics of endocrinology at two university hospitals and two general hospitals in the period from May 2010 to March 2012.
Pre-assignment Details: 163 patints screened. 44 screenfailures due to exclusion criteria as indicated. 119 randomized
Groups:
- Placebo: 1tablet of matching placebo trated up to 2 if neccessary
- Addition of Spironolactone: spironolactone is added to previous antihypertensive treatment
  placebo : addition of placebo 1 to 2 tablets daily
  spironolactone : 25 to 50 mg once daily
Period: Overall Study
Arm/Group | Placebo | Addition of Spironolactone
Started | 58 (119 randomized.) | 61
Completed | 55 | 57
Not Completed | 3 | 4
Not completed — Adverse Event | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Addition of Spironolactone | Placebo | Total
Number analyzed (Participants) | 61 | 58 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 28 | 62
  >=65 years | 27 | 30 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (7.1) | 63.9 (6.9) | 63.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 46 | 45 | 91
Region of Enrollment [Number; unit: participants]
  Denmark | 61 | 58 | 119

OUTCOME MEASURES:

1. Primary Outcome: Change of of Systolic Blood Pressure
Description: Change of systolic blood pressure from baseline to study end at four months.
Time Frame: 4 months
Population: Analysis by intention to treat using LOCF
Measure: Mean (95% Confidence Interval); unit: mm Hg
Groups:
- Addition of Spironolactone: spironolactone is added to previous antihypertensive treatment
  spironolactone : 25 uptrated if necessary to 50 mg once daily
- Placebo: 1tablet of matching placebo uptrated to 2 if neccessary
Arm/Group | Addition of Spironolactone | Placebo
Number analyzed (Participants) | 57 | 55
mm Hg | -9.6 [-12.8 to -6.3] | -0.7 [-3.3 to 2.0]

2. Secondary Outcome: Adverse Effects
Time Frame: 4 months
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Addition of Spironolactone | Placebo
Number analyzed (Participants) | 61 | 58
participants | 4 | 0

3. Primary Outcome: Change of Diastolic Blood Pressure
Description: Change of diastolic blood pressure from baseline to study end at four months.
Time Frame: 4 months
Population: Analyzed by intention to treat and last observation carried forward
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Addition of Spironolactone | Placebo
Number analyzed (Participants) | 57 | 55
mm Hg | -3.9 [-6.0 to -2.0] | -0.3 [-1.8 to 1.3]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Addition of Spironolactone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/61 | 0/58
Other Adverse Events (participants affected / at risk) | 0/61 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Addition of Spironolactone (N=61) | Placebo (N=58)
Serious hyperkalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Plasma potasium above 5.5 mmol/l

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No